CLINICAL TRIAL: NCT06377124
Title: A Smart Self-Management Support Programme (3S) to Improve Quality of Life in Patients With Lung Cancer - A Pragmatic Randomized Controlled Trial With Mixed-method Evaluation
Brief Title: A Smart Self-Management Support Programme (3S) to Improve Quality of Life in Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); The Queen Elizabeth Hospital (Other); United Christian Hospital (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Honorary Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW21-507
Record Dates: First submitted 2024-04-09; First posted 2024-04-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The 3S intervention includes an individual session, messaging and phone contact related to lung cancer self-management, and hotline services.
  The general health information includes an individual session, messaging and phone contact related to general health information, and hotline services.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was not aware of which groups the patients belonged to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The 3S intervention group (Experimental): Receive information and support on self-management of lung cancer
  Interventions: Behavioral: 3S intervention
- The GH information group (Placebo Comparator): Receive general health information such as sleep hygiene, environmental hygiene, etc.
  Interventions: Behavioral: GH information

INTERVENTIONS:
Behavioral: 3S intervention — The 3S intervention includes information and support related to self-management of lung cancer, including
  1. an individual 3S session at baseline,
  2. 24-week messaging, telephone coaching and hotline services.
  Arms: The 3S intervention group
Behavioral: GH information — The GH information includes information related to general health, including
  1. an individual GH session at baseline,
  2. 24-week messaging, telephone coaching and hotline services.
  Arms: The GH information group

SUMMARY:
Lung cancers patients often experience multiple symptoms (e.g. fatigue, dyspnea, distress, depression, sleep disturbance). The current study attempts to explore the efficacy of the Smart Self-Management Support Programme (3S) in improving quality of life of patients using self-management support programme with mobile devices.

DETAILED DESCRIPTION:
Lung cancer (LC) is the most and second most common cancer globally and locally respectively. LC patients often experience multiple symptoms (e.g. fatigue, dyspnea, distress, depression, sleep disturbance). The symptom burden is greater than other cancers and adversely affects quality of life. Care of LC patients has shifted from a purely disease-centered approach on survival-related outcomes to person-centered approach with emphasis on quality-of-life outcomes.

Self-management support programme (SMS) is perceived to supplement regular medical treatments and follow-up and cost-effective in cancer care. Besides, digital technologies have been used in patient empowerment digital platform to improve self-management of cancer patients. Using the self-management support programme and mobile devices, the Smart Self-Management Support Programme (3S) attempts to improve quality of life of patients.

The current study aims to examine the efficacy of 3S on improving quality of life and patient activation (knowledge, skills, and confidence for self-management) in the 3S intervention group, compared to the general health (GH) control group. It also aims to examine the changes in the burden of care, anxiety and depression symptoms, and quality of life of the family caregivers (FCGs) of the patients in the 3S group, compared to FCGs of the patients in the GH group.

We also conduct process valuations to assess the essential features of context, implementation, and impact mechanism, and cost-effectiveness evaluation to examine health care resource utilisation and cost-effectiveness analysis.

160 patients with lung cancer will be recruited, and 160 family caregivers will also be invited to join the study.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Aged 18 years or above
* Diagnosis of advanced-stage (stage III or stage IV) non-small cell lung cancer
* Ambulatory and capable of all self-care activities (ECOG ≤2)
* Either undergoing or has finished oncology therapy
* Mentally, cognitively and physically fit to join as determined by the doctor in charge and responsible clinical investigators
* Can speak and read Chinese
* Willing to complete the patient-reported outcome questionnaire
* Has a smartphone with WhatsApp or WeChat

Exclusion Criteria:

* Preparing for lung operation
* Skeletal fragility
* Serious active infection
* Inability to walk
* Previously untreated symptomatic brain metastases
* Severe respiratory insufficiency
* Uncontrolled pain
* Diagnosed psychiatric illness with or without medication

Family Caregivers:

Inclusion criteria:

* Aged 18 years or above
* Family caregivers of recruited patients

Exclusion criteria:

* Unable to speak and read Chinese
* Unwilling to complete the patient-reported outcome questionnaire

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life | Baseline and 8-week follow-up
  Measured by a 30-item European Organization for Research and Treatment of Cancer and Lung Module. All scale scores are linearly converted to a range from 0 to 100. Higher scores indicate better functioning and quality of life.

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline and 24-week follow-up
  Measured by a 30-item European Organization for Research and Treatment of Cancer and Lung Module. All scale scores are linearly converted to a range from 0 to 100. Higher scores indicate better functioning and quality of life.
Change in patient activation | Baseline, 8-week and 24-week follow-up
  Measured by a 13-item Patient Activation Measure with a 5-point Likert response scale from 0 to 4. Raw scores are transformed to a scale of 0-100 with higher scores indicating a higher activation in self-management.
Change in general self-efficacy | Baseline, 8-week and 24-week follow-up
  Measured by a 10-item General Self-efficacy Scale with a 4-point Likert response scale from 1 to 4, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Change in acceptance of illness | Baseline, 8-week and 24-week follow-up
  This is measured by a 12-item Peaceful Acceptance subscale of the Peace, Equanimity, and Acceptance in the Cancer Experience questionnaire. Each item ranges between 1 and 4. A higher score indicates a greater extent of acceptance of the cancer diagnosis.
Change in physical activity level | Baseline, 8-week and 24-week follow-up
  Measured the days and duration of physical activity level (light, moderate and vigorous) and sitting time in the past 7 days by the International Physical Activity Questionnaire (short version) with 4 questions.
Change in diet habit | Baseline, 8-week and 24-week follow-up
  Measured by 10-item dietary intake and practice outcome based questions
Change in smoking and drinking habits | Baseline, 8-week and 24-week follow-up
  Measured by self-reported drinking and smoking frequency
Change in health status | Baseline, 8-week and 24-week follow-up
  Measured by 5-item EuroQol-5D Questionnaire. Each item is a different dimension that ranges from level 1-5, a higher level indicates a more severe level of perceived problem of that dimension.
Change in anxiety symptoms of patients | Baseline, 8-week and 24-week follow-up
  Measured by a 7-item Generalised Anxiety Disorder Assessment. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 21. The higher scores the greater severity of anxiety symptoms.
Change in depression symptoms of patients | Baseline, 8-week and 24-week follow-up
  Measured by a 9-item Patient Health Questionnaire. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 27. The higher scores the greater severity of depression symptoms.
Change in social and family support | Baseline, 8-week and 24-week follow-up
  Measured by 8-item Family and Friend Subscales of Multidimensional Scale of Perceived Social Support with a 7-point Likert scale. Each scale ranges from 4 to 28. A higher score equates with higher social support.
Change in adherence to agreed preset health-related goals | Baseline, 8-week and 24-week follow-up
  Measured by web-based platform (WhatsApp) in which patients will be asked to self-report whether they have completed their previously agreed health-related or general hygiene goals with nurses on a weekly basis. Adherence will be assessed by the frequency of self-reported goal completion by patients.
Change in symptom severity | Baseline, 8-week and 24-week follow-up
  Measured by 13-item European Organization for Research and Treatment of Cancer on symptom severity with a 4-point Likert scale. A higher score indicates a higher level of symptom severity.
Change in functional exercise capacity | Baseline, 8-week and 24-week follow-up
  Measured by a 6-minute walk test. The distance of participant walked with the instructions to walk back and forth at their own pace to a designated spot for 6 minutes.
Change in lower limb strength | Baseline, 8-week and 24-week follow-up
  Measured by a 30-second chair stand test. The number of participant stood up repeatedly from a chair for 30 seconds.
Change in hand grip strength | Baseline, 8-week and 24-week follow-up
  Measured by a dynamometer
Change in flexibility | Baseline, 8-week and 24-week follow-up
  Measured by a Chair sit and reach test.
Change in balance | Baseline, 8-week and 24-week follow-up
  Measured by a single-leg stance test
Change in body composition | Baseline, 8-week and 24-week follow-up
  Calculated by ratio of body weight and body height
Change in objective physical activity level | Baseline, 8-week and 24-week follow-up
  Measured by a 7-day waist-worn accelerometer
Change in objective sleep quality | Baseline, 8-week and 24-week follow-up
  Measured by a sleep-wake monitor (Motionlogger MicroWatch)
Change in burden of family caregivers (For FCGs) | Baseline, 8-week and 24-week follow-up
  Measured by the 24-item Caregiver Burden Inventory with a 5-point Likert scale from 0 to 4. Total score ranges from 0 to 96 with higher score indicating a higher caregiver burden.
Change in quality of life of family caregivers (For FCGs) | Baseline, 8-week and 24-week follow-up
  Measured by the 35-item Caregiver Quality of Life Index-Cancer scale with a 5-point Likert scale from 0 to 4. Total score ranges from 0 to 140. Higher score indicates a higher quality of life.
Change in anxiety symptoms of family caregivers (For FCGs) | Baseline, 8-week and 24-week follow-up
  Measured by a 7-item Generalised Anxiety Disorder Assessment. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 21. The higher scores the greater severity of anxiety symptoms.
Change in depression symptoms of family caregivers (For FCGs) | Baseline, 8-week and 24-week follow-up
  Measured by a 9-item Patient Health Questionnaire. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 27. The higher scores the greater severity of depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Yuen Kwan Lai, PhD, Principal Investigator — School of Nursing and Health Sciences
Locations (3):
- Hong Kong (3):
  - Queen Elizabeth Hospital, Hong Kong, Ho ManTin
  - Queen Mary Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For those who want the patient data, please contact PI directly by written email.

REFERENCES:
- [Background] Kondylakis H, Bucur A, Crico C, Dong F, Graf N, Hoffman S, Koumakis L, Manenti A, Marias K, Mazzocco K, Pravettoni G, Renzi C, Schera F, Triberti S, Tsiknakis M, Kiefer S. Patient empowerment for cancer patients through a novel ICT infrastructure. J Biomed Inform. 2020 Jan;101:103342. doi: 10.1016/j.jbi.2019.103342. Epub 2019 Dec 6. PMID 31816400
- [Background] Saetan P, Chaiviboontham S, Pokpalagon P, Chansriwong P. The Effects of the Respiratory Rehabilitation Program on Perceived Self-Efficacy and Dyspnea in Patients with Lung Cancer. Asian Nurs Res (Korean Soc Nurs Sci). 2020 Dec;14(5):277-285. doi: 10.1016/j.anr.2020.08.010. Epub 2020 Sep 8. PMID 32916339
- [Background] Zhu X, Han S, Chu H, Wang M, Chen S. Influence of self-management exercise intervention on the cancer related fatigue severity and self-management efficacy of patients with non-small cell lung cancer after operation. J Pak Med Assoc. 2020 Sep;70 [Special Issue](9):88-93. PMID 33177734
- [Background] Hernandez Silva E, Lawler S, Langbecker D. The effectiveness of mHealth for self-management in improving pain, psychological distress, fatigue, and sleep in cancer survivors: a systematic review. J Cancer Surviv. 2019 Feb;13(1):97-107. doi: 10.1007/s11764-018-0730-8. Epub 2019 Jan 11. PMID 30635865
- [Background] Ji W, Kwon H, Lee S, Kim S, Hong JS, Park YR, Kim HR, Lee JC, Jung EJ, Kim D, Choi CM. Mobile Health Management Platform-Based Pulmonary Rehabilitation for Patients With Non-Small Cell Lung Cancer: Prospective Clinical Trial. JMIR Mhealth Uhealth. 2019 Jun 21;7(6):e12645. doi: 10.2196/12645. PMID 31228180